CLINICAL TRIAL: NCT06417138
Title: Comparative Effectiveness of Different Drugs Used to Treat Patients in Rheumatoid Arthritis Saudi Database (RASD) The Primary Objective of This Study is to Compare the Effectiveness of Different Biological Disease Modifying Antirheumatic Drugs (bDMARDs) and Targeted Synthetic (tsDMARDs) Using DAS-28-CRP and CDAI Scores.
Brief Title: Comparative Effectiveness of Different Drugs Used to tr€at Patients in Rheumatoid Arthritis Saudi Database (RASD)"
Status: Recruiting | Type: Observational
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Hani Mohammad Almoallim, Professor of Rheumatology, Umm Al-Qura University
Other Study IDs: 2023-0-225
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis RA
Keywords: Rheumatoid Arthritis; Remission; Biological DMARDs; Targeted synthetic DMARDs; DAS-28-CRP; CDAI; Low disease activity; Comparative effectiveness; Efficacy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis patients receiving biological DMARDs or targeted synthetic DMARDs: It will be a multicenter study. The data will be obtained primarily from Rheumatoid Arthritis Saudi Database (RASD). We will also include RA patients from other centers who are not part of the registry if they are providing minimum of 12 months follow up with at least 3 documented visits of these patients to health care facilities following "treat to target approach" or preferably "treat to work approach".
  Interventions: Other: biological and targeted synthetic disease modifying anti rheumatic drugs (bDMARDs) and (tsDMARDs)

INTERVENTIONS:
Other: biological and targeted synthetic disease modifying anti rheumatic drugs (bDMARDs) and (tsDMARDs) — This is a registry-based study. It is an observational, retrospective trial. There is/are no interventional drug(s).
  Other Names: bDMARDs; tsDMARDs

SUMMARY:
Comparative effectiveness of different drugs used to treat patients in Rheumatoid Arthritis Saudi database (RASD)

The goal of this observational study is to compare the effectiveness of different biological Disease Modifying Antirheumatic Drugs (bDMARDs) and targeted synthetic (tsDMARDs) using Disease Activity Score - 28 joints - C-Reactive Protien (DAS-28-CRP) and Clinical Disease Activity Index (CDAI) scores. In rheumatoid arthritis patients in Saudi Arabia who are part of Rheumatoid Arthritis Saudi Database (RASD).

The main question[s] it aims to answer:

* What is the most effective drug (biologocal or targeted synthetic) disease modifying antirheumatic drug used to treat rheumatoid arthritis in Saudi Arabia?
* We are going to use two outcome mesures: Disease Activity Score - 28 joints - C-Reactive Protien (DAS-28-CRP) and Clinical Disease Activity Index (CDAI) scores

Researchers will compare the treatment of rheumatoid arthritis using specific outcome measures in Rheumatoid Arthritis in Saudi Arabia.

* Participants will be enrolled after a signed written concent in our Rheumatoid Arthritis Saudi Databas (RASD).
* Their treatment data will used to compare the effectiveness of different drugs they are using.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic progressive inflammatory disease that causes irreversible joint deformities which can have debilitating effects on a patient's overall wellbeing. RA has a global prevalence rate of 0.5-1.1% with an annual incidence rate of 20-50 cases per 100 000 of the American and North European population.

Registries are widely mentioned in literature as a method that studied a given population in a way that is more applicable to clinical practice. Although there are numerous registries that previously set place in Europe and north America, the middle east and Africa remain scarcely studied with a few published small, scaled hospital reports. Registries are imperative to study a disease's unique course in each population, which may or may not align with its counterparts in western populations. Therefore, we established a Saudi registry for rheumatoid arthritis called Rheumatoid Arthritis Saudi Database (RASD).

We have published the results of RASD from one center recently. Our study was conducted in a single center in Saudi Arabia using a pool of 433 patients. The aim was to describe the population of rheumatoid arthritis and to compare these findings to previously published data registries.

Currently, RASD has expanded to include several centers in Saudi Arabia. It is essential to conduct a study that address the comparative effectiveness of different drugs used to treat RA in Saudi population. There are many reasons that make management of RA in our country different than other places in the world. This study should help us to compare our comparative effectiveness to other studies with similar methodologies that reported on effectiveness in different population than ours. We may include centers who are even not part of our RASD as long as they can provide a minimum of one year data on their RA patients with at least 3 visits describing the outcome measures that we are interested in.

By the end of this research project the following information will be available for health care leaders for strategic planning: The effectiveness of different biological and targeted synthetic DMARDs in Saudi population, showing the most effective and the least effective drug. This information can help in the following:

* Guide the development of a local guidelines focusing on the use of the most effective drugs in our population.
* Prioritizing the use of different drugs to treat RA in Saudi population.
* The drug survival rates and the discontinuation rates of different drugs in Saudi population.

This is a multicenter study. The data will be obtained primarily from Rheumatoid Arthritis Saudi Database (RASD). We will also include RA patients from other centers who are not part of the registry if they are providing minimum of 12 months follow up with at least 3 documented visits of these patients to health care facilities following "treat to target approach" or preferably "treat to work approach".

For the comparison of drug efficacy the best level of evidence is obtained by blinded randomized control design, however use of data of registry is also an acceptable option with known limitation. This is a retrospective study design. We will observe all the cohorts of registry as well as those meeting the criteria, to find out the most effective drug for the treatment of rheumatoid arthritis as well as to find out the association of various risk factors with the treatment outcome.

We will use non probability, convenience sampling technique to enroll the patients.

Sample size: Sample size was calculated as 798 based on a confidence interval of 95% and power of 80% with a p value of less than 0.05

All the collected data will be entered in SPSS version 22, edited, cleaned and analyzed. Categorical data will be measured by proportion and percentages while continuous data will be measured by mean and standard deviated where normality assumption is met. Homogeneity of variables will be measured by Levene's test for equality of variance. Student t test will be used to compare between two groups and ANOVA for the more than two groups in case of continuous data. For the categorical data Chi-Square test will be used for large data and Fisher Exact test for smaller data. Logistic regression model will be used in order to predict the outcome.

Exposure and outcome variables included: Age of patient, Age of onset, sex, urban vs rural areas, level of education, comorbidities, number of drugs used before using biological and targeted synthetic DMARDs, duration of methotrexate use before starting biological and targeted synthetic DMARDs, effectiveness of drugs, lag time, drug survival rate.

ELIGIBILITY:
Inclusion Criteria:

* All those patients who are age of 18 years and above and
* meeting 2010 American College of Rheumatology classification criteria for rheumatoid arthritis.
* Both male and female gender will be included.
* There should be minimum of 12 months follow up with at least 3 documented visits of these patients to health care facilities.

Exclusion Criteria:

* Any patient who did not meet the inclusion criteria will be excluded from the study.
* Any patient who cannot recall the exact date of starting his drugs will be excluded during data analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis patients who are enrolled in our rheumatoid arthritis Saudi Database will be included according the inclusion and exclusion criteria above. Other centers who are not part of RASD will be included as well as long as they will comply with study protocol and provide data as required.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
To compare the effectiveness of different biological Disease Modifying Antirheumatic Drugs (bDMARDs) and targeted synthetic (tsDMARDs) | "through study completion, an average of 1 year"
  using Disease Activity Score for 28 joints with C-Reactive Protein (DAS-28-CRP) (Remission <1.6, Low Disease Activity<2.4, Moderate Disease Activity<3.7, High Disease Activity >3.7)
To compare the effectiveness of different biological Disease Modifying Antirheumatic Drugs (bDMARDs) and targeted synthetic (tsDMARDs) | "through study completion, an average of 1 year"
  Using Clinical Disease Activity Index (CDAI) (Remission <2.8, Low Disease Activity <10, Moderate Disease Activity <22, High Disease Activity >22)

SECONDARY OUTCOMES:
Drug survival rate | "through study completion, an average of 1 year"
  The time that a specific drug has been used by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Hani Almoallim, Professor, Principal Investigator — Umm Al-Qura University
Locations (1):
- International medical center, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smolen JS, Landewe RBM, Bergstra SA, Kerschbaumer A, Sepriano A, Aletaha D, Caporali R, Edwards CJ, Hyrich KL, Pope JE, de Souza S, Stamm TA, Takeuchi T, Verschueren P, Winthrop KL, Balsa A, Bathon JM, Buch MH, Burmester GR, Buttgereit F, Cardiel MH, Chatzidionysiou K, Codreanu C, Cutolo M, den Broeder AA, El Aoufy K, Finckh A, Fonseca JE, Gottenberg JE, Haavardsholm EA, Iagnocco A, Lauper K, Li Z, McInnes IB, Mysler EF, Nash P, Poor G, Ristic GG, Rivellese F, Rubbert-Roth A, Schulze-Koops H, Stoilov N, Strangfeld A, van der Helm-van Mil A, van Duuren E, Vliet Vlieland TPM, Westhovens R, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2022 update. Ann Rheum Dis. 2023 Jan;82(1):3-18. doi: 10.1136/ard-2022-223356. Epub 2022 Nov 10. PMID 36357155
- [Background] Monti S, Montecucco C, Bugatti S, Caporali R. Rheumatoid arthritis treatment: the earlier the better to prevent joint damage. RMD Open. 2015 Aug 15;1(Suppl 1):e000057. doi: 10.1136/rmdopen-2015-000057. eCollection 2015. PMID 26557378
- [Background] Finckh A, Gilbert B, Hodkinson B, Bae SC, Thomas R, Deane KD, Alpizar-Rodriguez D, Lauper K. Global epidemiology of rheumatoid arthritis. Nat Rev Rheumatol. 2022 Oct;18(10):591-602. doi: 10.1038/s41584-022-00827-y. Epub 2022 Sep 6. PMID 36068354
- [Background] Almoallim H, Al Saleh J, Badsha H, Ahmed HM, Habjoka S, Menassa JA, El-Garf A. A Review of the Prevalence and Unmet Needs in the Management of Rheumatoid Arthritis in Africa and the Middle East. Rheumatol Ther. 2021 Mar;8(1):1-16. doi: 10.1007/s40744-020-00252-1. Epub 2020 Nov 23. PMID 33226566